CLINICAL TRIAL: NCT06420037
Title: The Influence of the Individual Auditory-cognitive Need on the Aided Benefit Using Different Feature Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: ONZ-2023-0437
Record Dates: First submitted 2024-04-16; First posted 2024-05-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Speech Intelligibility; Hearing Loss, Sensorineural
MeSH Terms: conditions — Speech Intelligibility; Hearing Loss, Sensorineural | interventions — Vision Screening; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individuals between 45-80 years with bilateral hearing aids (control group) (Other): Within this control group, no changes will be made to the hearing aid settings. However, they undergo all other tests of the test protocol.
  Interventions: Behavioral: Cognitive screening and vision screening; Behavioral: Audiological Assessment; Behavioral: Questionnaires; Behavioral: Cognition; Other: Real ear measurement
- Individuals between 45-80 years with bilateral hearing aids (frequency compression) (Experimental): Within this experimental group, a slight modification (which differs between groups) will be made to the basic hearing aid setting.
  Interventions: Device: Hearing aid feature adjustment (frequency compression) of the following hearing aids: Phonak Audéo Paradise/Lumity 70; Behavioral: Cognitive screening and vision screening; Behavioral: Audiological Assessment; Behavioral: Questionnaires; Behavioral: Cognition; Other: Real ear measurement
- Individuals between 45-80 years with bilateral hearing aids (noise reduction) (Experimental): Within this experimental group, a slight modification (which differs between groups) will be made to the basic hearing aid setting.
  Interventions: Device: Hearing aid feature adjustment (noise reduction) of the following hearing aids: Phonak Audéo Paradise/Lumity 70; Behavioral: Cognitive screening and vision screening; Behavioral: Audiological Assessment; Behavioral: Questionnaires; Behavioral: Cognition; Other: Real ear measurement

INTERVENTIONS:
Device: Hearing aid feature adjustment (frequency compression) of the following hearing aids: Phonak Audéo Paradise/Lumity 70 — Upon enrollment, each participant will be allocated to one of three research groups and participants will remain unaware of their group assignment. This groups will undergo a slight modification, namely frequency compression turned off, to the basic setting.
  Arms: Individuals between 45-80 years with bilateral hearing aids (frequency compression)
Device: Hearing aid feature adjustment (noise reduction) of the following hearing aids: Phonak Audéo Paradise/Lumity 70 — Upon enrollment, each participant will be allocated to one of three research groups and participants will remain unaware of their group assignment. This groups will undergo a slight modification, namely noise reduction turned off, to the basic setting.
  Arms: Individuals between 45-80 years with bilateral hearing aids (noise reduction)
Behavioral: Cognitive screening and vision screening — The Dutch Montreal Cognitive Assessment will be assessed. The Snellen Eye Test will be used to screen for normal or corrected-to-normal vision.
Behavioral: Audiological Assessment — Three audiological tests are included: 1) Tympanometry to assess the middle ear status, 2) Pure-tone audiometry with headphone to evaluate the hearing thresholds, 3) Speech audiometry in free field to assess the ability to understand spoken sentences in quiet and in the presence of background noise.
Behavioral: Questionnaires — Three questionnaires are included:
  1. The HAVICOP questionnaire to assess the hearing-related quality of life (Ceuleers, D., Baudonck, N., Keppler, H., Kestens, K., Dhooge, I., & Degeest, S. (2023). Development of the hearing-related quality of life questionnaire for auditory-visual, cognitive and psychosocial functioning (hAVICOP). Journal of communication disorders, 101, 106291.)
  2. the FAS (fatigue assessment scale) to assess how you usually feel
  3. the EEAS (extended effort assessment scale) to assess how you experience listening in everyday life.
Behavioral: Cognition — Four cognitive functions, important for speech understanding, will be assessed both audibly and visually: divided attention, working memory, processing speed, and cognitive flexibility and inhibition.
Other: Real ear measurement — This test will give an objective assessment of the hearing aids' configuration.

SUMMARY:
The goal of this clinical trial is to optimize hearing aid benefit based on the individual auditory-cognitive need using different hearing aid features in first-time hearing aid users between 45-80 years old with bilateral Phonak Audéo Paradise/Lumity 70/90 hearing aids. The main questions it aims to answer are:

Does cognitive functioning affect hearing aid benefit? How can hearing aid fitting be optimized based on the individual auditory-cognitive profile?

The hypothesis posits that cognitive abilities influence the effectiveness of hearing aids, alongside hearing status. Furthermore, if features of hearing aids improve speech understanding and listening effort, it is proposed that individuals with lower cognitive functioning will experience heightened benefits from hearing aids.

The study will consist of three groups: one control group and two groups where one different feature will be modified.

Participants will be tested at baseline measurement, including:

* screening tests
* audiological tests
* questionnaires
* cognitive tests
* real-ear-measurement

Following this, participants will be divided in one of the three groups, after which speech audiometry will be repeated. After a 4-week acclimatization period, the second measurement will take place, repeating speech audiometry and questionnaires. Subsequently, the hearing aid settings will be restored to their initial configuration.

ELIGIBILITY:
Inclusion Criteria:

* Dutch-speaking individuals aged between 45-80 years old
* individuals with normal vision (with glasses or lenses if needed)
* individuals with age-related hearing loss
* individuals with bilateral hearing aids (Phonak Audéo Paradise/Lumity 70)
* individuals who are capable to give consent to participate in the study themselves

Exclusion Criteria:

* user of cochlear implants
* use of influencing medication (for example: Rilatin and antidepressants)
* learning disabilities (for example: dyslexia and dyscalculia)
* (history of) neurological problems (brain tumor, epilepsy, history of stroke, ...)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Speech reception threshold | This outcome measure will be assessed twice during the initial measurement (both +/- 10 minutes) and once during the second measurement (+/- 10 minutes).
  Based on the results of the speech understanding task, the speech reception threshold will give an indication of the ability to understand spoken sentences in quiet and noise.

SECONDARY OUTCOMES:
Hearing related quality of life | This outcome parameter will be assessed twice: once during the initial measurement and once during the subsequent measurement (both +/- 10 minutes).
  Thirty-five sentences should be responded using a VAS (0-100). Mean scores will be calculated for each subdomain separately (auditory-visual, cognitive, and psychosocial functioning) as well as combined within a total score; the worse one's hearing-related quality of life, the lower the score.
Fatigue assessment | This outcome parameter will be assessed twice: once during the initial measurement and once during the subsequent measurement (both +/- 5 minutes).
  Ten sentences should be responded based on five categories, ranging from Never to Always: 1 = Never; 2 = Sometimes; 3 = Frequently; 4 = Often; and 5 = Always.
Effort assessment | This outcome parameter will be assessed twice: once during the initial measurement and once during the subsequent measurement (both +/- 5 minutes).
  Ten sentences should be responded using a VAS (0-100). Mean scores will be calculated for each sentence. The lower the score, the lower the effort.
Cognitive functioning (auditory and visual) | These outcome measures will be assessed once during the first measurement (+/- 55 minutes).
  Cognitive functions such as 'divided attention', 'working memory', 'processing speed', and 'flexibility and inhibition' will be assessed both audibly and visually. Mean scores and average reaction times will be computed.
Real ear measurement | This outcome measure will be assessed once during the first measurement (+/- 15-20 minutes).
  Test to obtain an objective understanding of the current settings of the hearing aids.
Screening of mild cognitive impairment (MoCA) and vision | This outcome measure will be assessed once during the first measurement (+/- 5-10 minutes).
  The result (max 30) on the MoCA will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Keppler, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, East-Flanders, Belgium